CLINICAL TRIAL: NCT05745064
Title: A Phase 2, Multicenter, Randomized, Double-masked, Placebo-controlled Study to Evaluate the Safety and Tolerability of TL-925 Ophthalmic Emulsion 0.1% in Subjects With Moderate to Severe Dry Eye Disease
Brief Title: A Study of TL-925 as a Treatment for Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TL-925-301
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Disease
Keywords: TL-925; Phase II
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: In this prospective, Phase 2, multicenter, randomized, double-masked, placebo-controlled, parallel-arm study, approximately 100 subjects with moderate to severe dry eye disease (DED) will be randomly assigned (1:1) to receive either TL-925 or placebo as topical ophthalmic eye drops administered bilaterally BID.
  The study will comprise two phases: 2-weeks screening/run-in and 4-weeks double-masked treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor, Investigators and study staff will be masked during the randomization process and throughout the study. The study site will have the capacity to unmask participants in an emergency.
  Following completion of the study, the randomization code will be unmasked once all data has been entered into the Study database for every subject and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TL-925 Arm (Active Comparator): TL-925 will be administered OU BID
  Interventions: Drug: TL-925
- Placebo Arm (Placebo Comparator): Placebo will be administered OU BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TL-925 — TL-925 is an eye drop.
  Arms: TL-925 Arm
Drug: Placebo — The composition of the placebo is identical to the active formulation except for the exclusion of the active ingredient.
  Arms: Placebo Arm

SUMMARY:
In this prospective, Phase 2, multicenter, randomized, double-masked, placebo-controlled, parallel-arm study, approximately 100 subjects with moderate to severe dry eye disease (DED) will be randomly assigned (1:1) to receive either TL-925 or placebo as topical ophthalmic eye drops administered bilaterally BID.

The study will comprise two phases: 2-weeks screening/run-in and 4-weeks double-masked treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* A diagnosis of dry eye disease for at least 6 months
* An unanesthetized Schirmer's test score (STS) of ≤ 10mm and ≥ 1mm in the study eye
* A tear film break-up time (TFBUT) of ≤ 5 seconds in the study eye
* A corneal fluorescein staining score of ≥ 2 in at least one region of the cornea
* A sum corneal fluorescein staining score of ≥ 4 in the study eye
* A total lissamine green conjunctival score of ≥ 2 in the study eye
* Female subjects of childbearing potential and their male partners must both use a highly effective contraception method during the study.

Exclusion Criteria:

* Any clinically significant slit lamp finding
* Any ongoing ocular infection (bacterial, viral or fungal) or active ocular inflammation
* Any keratorefractive surgery within the last 12 months
* Any intraocular or extraocular surgery within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Adverse events during screening & treatment period | Baseline to the end of day 29 (±2 days)

SECONDARY OUTCOMES:
Change from baseline in corneal and conjunctival staining | Baseline to the end of day 29 (±2 days)
  Fluorescein staining by region in designated study eye will be used. Results will be assessed using a 5-point Corneal and Conjunctival Staining Scale.
Change from baseline in ocular discomfort | Baseline to the end of day 29 (±2 days)
  Visual analog scale (VAS) will be used. This will assess patients on a a 7-item 100-point scale based on ocular discomfort.
Change from baseline visual acuity | Baseline to the end of day 29 (±2 days)
  Best corrected visual acuity (BCVA) will be used to determine change in visual acuity from baseline.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Aesthetic Eye Care, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Michael Washburn Center for Ophthalmic Research, LLC., Indianapolis, Indiana
  - Andover Eye Associates, Andover, Massachusetts